CLINICAL TRIAL: NCT03721653
Title: Randomized Phase II Study of FOLFOXIRI Plus Bevacizumab Plus Atezolizumab Versus FOLFOXIRI Plus Bevacizumab as First-line Treatment of Unresectable Metastatic Colorectal Cancer Patients.
Brief Title: FOLFOXIRI + Bev + Atezo vs FOLFOXIRI + Bev as First-line Treatment of Unresectable Metastatic Colorectal Cancer Patients
Acronym: AtezoTRIBE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gruppo Oncologico del Nord-Ovest (Other)
Collaborators: Roche Pharma AG (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-000977-35
Record Dates: First submitted 2018-10-25; First posted 2018-10-26 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Metastatic Colorectal Cancer
Keywords: FOLFOXIRI; Bevacizumab; Atezolizumab
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Irinotecan; Oxaliplatin; Leucovorin; Fluorouracil; atezolizumab

STUDY DESIGN:
Intervention Model Description: prospective, open-label, multicentric phase II randomized in a 1:2 ratio
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FOLFOXIRI + Bevacizumab (Active Comparator): (to be repeated every 2 weeks for a maximum of 8 cycles) Bevacizumab 5 mg/kg iv over 30 minutes day 1, followed by Irinotecan 165 mg/sqm iv over 60 minutes day 1, followed by Oxaliplatin 85 mg/sqm iv over 2 hours day 1, in two-way with L-Leucovorin 200 mg/sqm iv over 2 hours day 1, followed by 5-fluorouracil 3200 mg/sqm 48 h-continuous infusion, starting on day 1 (to be repeated every 2 weeks for a maximum of 8 cycles)
  If no progression occurs during FOLFOXIRI plus bev, patients will receive maintenance 5-FU/LV plus bev at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus bev will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  The prosecution of bev until disease progression is recommended also if 5-FU is interrupted because of adverse events, patient's refusal or investigator's choice.
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: L-Leucovorin; Drug: 5-fluorouracil
- FOLFOXIRI + Bevacizumab + Atezolizumab (Experimental): Atezolizumab 840 mg iv over 30 minutes(60 minutes at the first infusion) day 1 followed by Bevacizumab 5 mg/kg iv over 30 minutes day 1, followed by Irinotecan 165 mg/sqm iv over 60 minutes day 1, followed by Oxaliplatin 85 mg/sqm iv over 2 hours day 1, in two-way with L-Leucovorin 200 mg/sqm iv over 2 hours day 1, followed by 5-fluorouracil 3200 mg/sqm 48 h-continuous infusion, starting on day 1 (to be repeated every 2 weeks for a maximum of 8 cycles)
  If no progression occurs during FOLFOXIRI plus bev plus atezolizumab, patients will receive maintenance 5-FU/LV plus bev plus atezolizumab at the same dose used at the last cycle of the induction treatment. 5-FU/LV plus bev plus atezolizumab will be repeated biweekly until disease progression, unacceptable toxicity or patient's refusal.
  The prosecution of bev and atezolizumab until disease progression is recommended also if 5-FU is interrupted because of adverse events, patient's refusal or investigator's choice.
  Interventions: Drug: Bevacizumab; Drug: Irinotecan; Drug: Oxaliplatin; Drug: L-Leucovorin; Drug: 5-fluorouracil; Drug: Atezolizumab

INTERVENTIONS:
Drug: Bevacizumab — 5 mg/kg iv over 30 minutes day 1
Drug: Irinotecan — 165 mg/sqm iv over 60 minutes day 1
Drug: Oxaliplatin — 85 mg/sqm iv over 2 hours day 1
Drug: L-Leucovorin — 200 mg/sqm iv over 2 hours day 1
Drug: 5-fluorouracil — 3200 mg/sqm 48 h-continuous infusion
Drug: Atezolizumab — 840 mg iv over 30 minutes (60 minutes at the first infusion) day 1
  Arms: FOLFOXIRI + Bevacizumab + Atezolizumab

SUMMARY:
The scope of this study is to evaluate the efficacy of the addition of atezolizumab to FOLFOXIRI plus bevacizumab as first line treatment of patients with metastatic colorectal cancer in terms of Progression Free Survival.

DETAILED DESCRIPTION:
This is a prospective, open-label, multicentric phase II randomized in a 1:2 ratio trial in which patients initially unresectable and previously untreated mCRC will receive induction treatment with FOLFOXIRI plus bev up to 8 cycles followed by maintenance with 5-FU/LV plus bev until disease progression, unacceptable toxicity or patient's refusal (arm A) versus FOLFOXIRI plus bev plus atezolizumab up to 8 cycles followed by maintenance with 5-FU/LV plus bev plus atezolizumab until disease progression, unacceptable toxicity or patient's refusal (arm B). If disease progression does not occur during induction, at the treating physician's discretion, the reintroduction after progression of the same induction treatment (up to 8 cycles) according to randomization arm, followed by maintenance until disease progression, unacceptable toxicity or patient's refusal, is recommended.

The third- and subsequent lines of treatment will be at investigators' choice.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent to study procedures
* Histologically proven diagnosis of colorectal cancer
* Initially unresectable metastatic colorectal cancer not previously treated with chemotherapy for metastatic disease
* At least one measurable lesion according to RECIST1.1 criteria
* Availability of a tumoral sample
* Male or female of 18-75 years of age
* ECOG PS < or = 2 if aged < 71 years, ECOG PS = 0 if aged 71-75 years
* Life expectancy of at least 12 weeks
* Previous adjuvant chemotherapy allowed only if with fluoropyrimidine monotherapy and more than 6 months elapsed between the end of adjuvant and first relapse
* Neutrophils >1.5 x 109/L, Platelets >100 x 109/L, Hgb >9 g/dl
* Total bilirubin 1.5 time the upper-normal limits (UNL) of the normal values and ASAT (SGOT) and/or ALAT (SGPT) <2.5 x UNL (or <5 x UNL in case of liver metastases) alkaline phosphatase <2.5 x UNL (or <5 x UNL in case of liver metastases)
* Creatinine clearance ≥50 mL/min or serum creatinine 1.25 x UNL
* INR or aPTT ≤1.5 × ULN. Patients who are on therapeutic doses of anti-coagulants are eligible if they are on a stable dose of anti-coagulant for 28 days with stable INR and PTT values
* Urine dipstick of proteinuria <2+. Patients discovered to have 2+ proteinuria on dipstick urinalysis at baseline, should undergo a 24-hour urine collection and must demonstrate ≤1 g of protein/24 hr
* Male subjects with female partners of childbearing potential must be willing to use adequate contraception as outlined in Section 5.5 - Contraception, starting with the first dose of study therapy through 6 months after the last dose of bevacizumab and within 5 months after the last dose of atezolizumab.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

* Women of childbearing potential must have a negative blood pregnancy test at the baseline visit. For this trial, women of childbearing potential are defined as all women after puberty, unless they are postmenopausal for at least 12 continuous months, are surgically sterile, or are sexually inactive.
* Female subjects of childbearing potential must be willing to use an adequate method of contraception as outlined in Section 5.5 - Contraception, for the course of the study starting with the first dose of study therapy through 6 months after the last dose of bevacizumab and within 5 months after the last dose of atezolizumab.

Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject

• Will and ability to comply with the protocol

Exclusion Criteria:

* Radiotherapy to any site within 4 weeks before the study
* Previous adjuvant oxaliplatin-containing chemotherapy
* Previous treatment with bevacizumab
* Prior treatment with CD137 agonists, anti-CTLA4, anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Untreated brain metastases or spinal cord compression or primary brain tumours
* History or evidence upon physical examination of CNS disease unless adequately treated
* Hystory of haemoptysis ≥2 grade NCIC-CTG criteria within one month prior screening
* Active or untreated CNS metastases. Patients with a history of treated asymptomatic CNS metastases are eligible provided they meet all the following criteria:
* Measurable disease outside the CNS
* Only supratentorial or cerebellar metastases allowed (i.e. no metastases to midbrain, pons, medulla or spinal cord)
* No ongoing requirement for corticosteroid therapy for CNS disease
* Symptomatic peripheral neuropathy > 2 grade NCIC-CTG criteria
* Serious, non-healing wound, ulcer, or bone fracture
* Evidence of bleeding diathesis or coagulopathy
* Uncontrolled hypertension and prior histor of hypertensive crisis or hypertensive encephalopathy
* Clinically significant (i.e. active) cardiovascular disease for example cerebrovascular accidents (≤6 months), myocardial infarction (≤6 months), unstable angina, New York Heart Association (NYHA) grade II or greater congestive heart failure, serious cardiac arrhythmia requiring medication
* Significant vascular disease (e.g. aortic aneurysm requiring surgical repair or recent arterial thrombosis) within 6 months of study enrolment.
* Active infection requiring antibiotics at the time of initiation of study treatment.
* Any previous venous thromboembolism ≥ NCI CTCAE Grade 4.
* History of abdominal fistula, GI perforation, intra-abdominal abscess or active GI bleeding within 6 months prior to the first study treatment.
* Current or recent (within 10 days prior to study treatment start) ongoing treatment with anticoagulants for therapeutic purposes
* Chronic, daily treatment with high-dose aspirin (>325 mg/day)
* Treatment with any investigational drug within 30 days prior to enrollment or 2 investigational agent half-lives (whichever is longer)
* Other co-existing malignancies or malignancies diagnosed within the last 5 years with the exception of localized basal and squamous cell carcinoma or cervical cancer in situ
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to study treatment start, or anticipation of the need for major surgical procedure during the course of the study
* Core biopsy or other minor surgical procedure, excluding placement of a vascular access device, within 7 days prior to initiation of study treatment
* Lack of physical integrity of the upper gastrointestinal tract, malabsorption syndrome, or inability to take oral medication
* Pregnant or lactating women. Women of childbearing potential with either a positive or no pregnancy test at baseline. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Sexually active males and females (of childbearing potential) unwilling to practice contraception (barriere contraceptive measure or oral contraception) during the study and until 6 months after the last dose of bevacizumab and within 5 months after the last dose of atezolizumab.
* History of autoimmune disease including but not limited to myasthenia gravis, myositis, autoimmune hepatitis, systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, vascular thrombosis associated with antiphospholipid syndrome, Wegener's granulomatosis, Sjögren's syndrome, Guillain-Barré syndrome, multiple sclerosis, vasculitis, or glomerulonephritis.

Note: History of autoimmune-related hypothyroidism on a stable dose of thyroid replacement hormone may be eligible for this study.

Note: Controlled Type 1 diabetes mellitus on a stable insulin regimen may be eligible for this study.

* History of idiopathic pulmonary fibrosis (including pneumonitis), drug-induced pneumonitis, organizing pneumonia (i.e., bronchiolitis obliterans, cryptogenic organizing pneumonia), or evidence of active pneumonitis on screening chest CT scan Note: History of radiation pneumonitis in the radiation field (fibrosis) is permitted
* Positive test for human immunodeficiency virus (HIV)
* Active hepatitis B (defined as having a positive hepatitis B surface antigen [HBsAg] test prior to randomization) or hepatitis C Note: Patients with past hepatitis B virus (HBV) infection or resolved HBV infection (defined as having a negative HBsAg test and a positive antibody to hepatitis B core antigen [anti-HBc] antibody test) are eligible.

Note: Patients positive for hepatitis C virus (HCV) antibody are eligible only if polymerase chain reaction (PCR) is negative for HCV RNA.

* Active tuberculosis
* Prior allogenic bone marrow transplantation or solid organ transplant
* Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumour necrosis factor [TNF] agents) within 2 weeks prior to start of study treatment, or requirement for systemic immunosuppressive medications during the trial. The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.

Note: Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the study.

* Known hypersensitivity or allergy to Chinese hamster ovary cell products or any component of the atezolizumab formulation
* Administration of a live, attenuated vaccine within 4 weeks prior to start of study treatment or anticipation that such a live attenuated vaccine will be required during the study
* Treatment with systemic immunostimulatory agents (including but not limited to interferons or interleukin-2) within 4 weeks or five half-lives of the drug, whichever is longer, prior to start of study treatment
* If receiving a RANKL inhibitor (e.g. denosumab), unwilling to adopt alternative treatment such as (but not limited to) bisphosphonates, while receiving atezolizumab.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 218 (Actual)
Dates: Start 2018-11-30 (Actual); Primary Completion 2021-06-15 (Actual); Study Completion 2023-08-31 (Actual)

PRIMARY OUTCOMES:
Progression Free Survival (PFS) | 16 months
  Progression-free survival is defined as the time from randomization to the first documentation of objective disease progression or death due to any cause, whichever occurs first.

SECONDARY OUTCOMES:
Overall toxicity rate | 24 months
  Overal Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing any adverse event, according to National Cancer Institute Common Toxicity Criteria (version 4.0), during the induction and the maintenance phases of treatment.
Toxicity rate | 24 months
  Toxicity Rate is defined as the percentage of patients, relative to the total of enrolled subjects, experiencing a specific adverse event of grade 3/4, according to National Cancer Institute Common Toxicity Criteria (version 4.0), during the induction and the maintenance phases of treatment.
Objective response rate according to RECIST version 1.1 criteria (ORR) | 16 months
  Objective Response Rate (ORR) is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to RECIST 1.1 criteria, during the induction and the maintenance phases of treatment. The determination of clinical response will be based on investigator reported measurements. Responses will be evaluated every 8 weeks.
Immuno-related objective response rate according to modified RECIST criteria (irORR) | 16 months
  Immuno-related Objective Response Rate (irORR) is defined as the percentage of patients, relative to the total of enrolled subjects, achieving a complete (CR) or partial (PR) response, according to immune-modified RECIST criteria, during the induction and the maintenance phases of treatment. The determination of clinical response will be based on investigator reported measurements. Responses will be evaluated every 8 weeks.
Early Objective Response Rate (EOR) | 16 months
  Early Objective Response Rate (EOR) is defined as the percentage of patients, relative to the total of the enrolled subjects, achieving a ≥ 20% decrease in the sum of diameters of RECIST target lesions at week 8 compared to baseline.
Deepness of response (DoR) | 16 months
  Deepness of Response (DoR) is defined as the relative change in the sum of longest diameters of RECIST target lesions at the nadir, in the absence of new lesions or progression of non-target lesions, when compared with baseline.
R0 Resection Rate | 16 months
  R0 Resection Rate is defined as the percentage of patients, relative to the total of enrolled subjects, undergoing secondary R0 resection of metastases. Secondary R0 surgery is defined as microscopically margin free complete surgical removal of all residual disease, performed during treatment or after its completion, allowed by tumoral shrinkage and/or disappearance of one or more lesions.
Progression Free Survival 2 (PFS2) | 18 months
  Progression Free Survival 2 (PFS2) is defined as beginning with randomization and ending with the first of the following events: a) death; b) disease progression according to RECIST 1.1 criteria on any treatment given after 1st progression. For patients that will not receive any treatment within 3 months after 1st progression, PFS2 will be equal to PFS. Censoring rules for PFS2 will be: end of study without PD, loss at follow-up. Curative surgery for metastasis will not result in censoring for PFS2.
  PFS2 will be analyzed both in the intention-to-treat population (whichever 2nd-line treatment will be adopted) and in the per-protocol population.
2nd-PFS | 18 months
  2nd-Progression free survival (2nd-PFS) is defined as the time from the beginning of the second-line treatment to the documentation of objective disease progression according to RECIST 1.1 criteria or death due to any cause, whichever occurs first. 2nd-PFS will be censored on the date of the last evaluable on study tumor assessment documenting absence of progressive disease for patients who are alive, on study and 2nd-progression free at the time of the analysis. 2nd-PFS will be analyzed both in the intention-to-treat population (whichever 2nd-line treatment will be adopted) and in the per-protocol population.

CONTACTS AND LOCATIONS:
Locations (1):
- Francesca Vannini, Pisa, Italia, Italy

REFERENCES:
- [Derived] Antoniotti C, Rossini D, Pietrantonio F, Salvatore L, Lonardi S, Tamberi S, Marmorino F, Moretto R, Prisciandaro M, Tamburini E, Tortora G, Passardi A, Bergamo F, Raimondi A, Ritorto G, Borelli B, Conca V, Ugolini C, Aprile G, Antonuzzo L, Gelsomino F, Martinelli E, Pella N, Masi G, Boni L, Galon J, Cremolini C. Upfront Fluorouracil, Leucovorin, Oxaliplatin, and Irinotecan Plus Bevacizumab With or Without Atezolizumab for Patients With Metastatic Colorectal Cancer: Updated and Overall Survival Results of the ATEZOTRIBE Study. J Clin Oncol. 2024 Aug 1;42(22):2637-2644. doi: 10.1200/JCO.23.02728. Epub 2024 Jun 12. PMID 38865678
- [Derived] Antoniotti C, Rossini D, Pietrantonio F, Catteau A, Salvatore L, Lonardi S, Boquet I, Tamberi S, Marmorino F, Moretto R, Ambrosini M, Tamburini E, Tortora G, Passardi A, Bergamo F, Kassambara A, Sbarrato T, Morano F, Ritorto G, Borelli B, Boccaccino A, Conca V, Giordano M, Ugolini C, Fieschi J, Papadopulos A, Massoue C, Aprile G, Antonuzzo L, Gelsomino F, Martinelli E, Pella N, Masi G, Fontanini G, Boni L, Galon J, Cremolini C; GONO Foundation Investigators. Upfront FOLFOXIRI plus bevacizumab with or without atezolizumab in the treatment of patients with metastatic colorectal cancer (AtezoTRIBE): a multicentre, open-label, randomised, controlled, phase 2 trial. Lancet Oncol. 2022 Jul;23(7):876-887. doi: 10.1016/S1470-2045(22)00274-1. Epub 2022 May 27. PMID 35636444
- [Derived] Antoniotti C, Borelli B, Rossini D, Pietrantonio F, Morano F, Salvatore L, Lonardi S, Marmorino F, Tamberi S, Corallo S, Tortora G, Bergamo F, Brunella DS, Boccaccino A, Grassi E, Racca P, Tamburini E, Aprile G, Moretto R, Boni L, Falcone A, Cremolini C. AtezoTRIBE: a randomised phase II study of FOLFOXIRI plus bevacizumab alone or in combination with atezolizumab as initial therapy for patients with unresectable metastatic colorectal cancer. BMC Cancer. 2020 Jul 22;20(1):683. doi: 10.1186/s12885-020-07169-6. PMID 32698790